CLINICAL TRIAL: NCT06923163
Title: Metabolic Response of Sedentary Participants to a Long-term Exercise Intervention
Brief Title: The Effect of Exercise on Metabolic Alteration
Acronym: Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIAT-IRB-240615-H0892; SIATCAS (Registry Identifier: Shenzhen Institutes of Advanced Technology，Chinese Academy of Sciences)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Behavior; Healthy Participants; Adult
Keywords: Metabolic response; Energy expenditure; Energy compensation
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental): Participants will run on treadmill under the supervision of the researcher
  * Intensity:60% of VO2max
  * Duration: for 12 weeks
  * Frequency: 5 times a week.
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — Exercise prescription for participant，
  * 150Kcal for Weeks 1-4 (gradually increase to 150Kcal in the first two weeks as familiar stage),
  * 250Kcal for Weeks 5-8,
  * 350Kcal for Weeks 9-12.
  Other Names: physical activity

SUMMARY:
The goal of this clinical trial is to study the effectiveness of aerobic exercise in treating obesity in adults and to assess the efficacy of exercise. The primary research questions it seeks to address are as follows:

* To what extent does exercise increase the total energy expenditure of participants?
* Why and how does the energy expenditure from exercise not fully compensate for the total energy expenditure (TEE)?
* Researchers will assess the efficacy and potential challenges of using exercise as a treatment for obesity by comparing the measurement data before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).

Participants will engage in the following activities:

* Engage in running sessions supervised five times a week for a duration of 12 weeks.
* Attend laboratory sessions both before and after the exercise intervention period for metabolic and anthropometric measurements, as well as sample collection.
* Return to the laboratory for further metabolic and anthropometric measurements and sample collection8 weeks post-completion of exercise intervention.

DETAILED DESCRIPTION:
Based on previous research findings, scientists found that exercise results in energy compensation. In a non-interventional setting, energy intake and expenditure undergo a dynamic equilibrium process. Nonetheless, the energy deficit induced by exercise is offset by other physiological or psychological behaviors, leading to a diminished energy discrepancy caused by exercise, thereby mitigating the weight loss effects typically associated with exercise(Pontzer et al 2016: Current Biology).Controlled dietary experiments have indicated that long-term exercise results in approximately 22% energy compensation (Bouchard et al 1994: Obesity Research); however, the underlying source and mechanism of this compensation remains ambiguous. Analyses of Total Energy Expenditure (TEE) in 1754 individuals have demonstrated that the energy compensation from exercise primarily emanates from a reduction in Basal Energy Expenditure (BEE), with only an average of 72% of the energy expended during exercise being utilized for additional energy expenditure (Careau et al 2021: Current Biology). Nevertheless, this deduction is restricted by the measurements of energy intake, Adaptive thermogenesis, Thermic Effect of Food (TEF), and Activity-related Energy Expenditure (AEE), emphasizing the necessity of exercise intervention studies to comprehensively grasp the pathways and mechanisms of energy compensation.

To tackle the challenges posed by overweight and obesity, enhance residents' quality of life, and delve deeper into the intricacies of energy compensation, this research project focuses on examining the metabolic reactions of the body to exercise interventions. Through the analysis of pre- and post-exercise energy expenditure and intake, body composition, metabolism, microbiota, and metabolomics alterations in humans, the primary goal is to thoroughly elucidate the principal factors and mechanisms behind energy compensation. This clinical trial consists of four phases: pre-exercise intervention baseline measurement, exercise intervention, Immediately after 12 weeks' exercise intervention measurement, and follow-up measurement 8 weeks post-completion of the exercise intervention.

Pre-exercise intervention baseline measurement:

* Anthropometric measurements: body weight, height, and body composition

  * Body weight: At visit 1, fasting body weight will be measured using a calibrated seca at the beginning of the visit. Fasting weight will be measured at visit 2 and, if applicable.
  * Height: Height (to +0.1 cm) will be measured by seca 217 stable without wearing shoes.
  * Body composition:

    * Fat mass will be measured by Magnetic Resonance Imaging (MRI, Shanghai united imaging, uMR 790 ).
    * Bioimpedance analysis will measure fat-free mass (Tanita, MC-980).
    * Bone mass will be measured by Dual Energy X-ray Absorptiometry (DXA, Horizon Wi, HOLOGIC).
* Metabolic measurements: blood pressure, glucose, heart rate, energy expenditure, and cardiovascular function

  * Blood pressure： Systolic and diastolic blood pressure will be measured using an Omron digital sphygmomanometer.
  * Blood glucose： Fasting and post-prandial glucose will be recorded by a continuous glucose monitoring system.
  * Heart rate：Heart rate will be monitored by a continuous heart rate monitoring system.
  * Energy expenditure：

    * TEE will be measured using the doubly-labeled water (DLW) method. Urine samples from all participants in the DLW subset will be stored at -20℃ and shipped on dry ice for analysis in the laboratory of Prof. John Speakman at the Shenzhen Institutes of Advanced Technology, Chinese academy of sciences. Isotopes will be measured in benchtop near-infrared isotope gas analyzer, and mean CO2 production will be calculated from isotope ratios using the recently derived equation (Speakman et al 2021: Cell reports medicine). TEE will then be calculated using mean CO2 production.
    * Resting Energy Expenditure (REE) and TEF will be measured by indirect calorimetry while participants are resting supine in a respiratory chamber with thermoneutral conditions. Oxygen consumption and CO2 production will be measured to calculate energy expenditure. REE will be consistently measured throughout sleeping at night and in the morning after overnight fasting, and TEF will be measured after breakfast.
  * VO2max test：Participants must warm up with simple stretching or light aerobic exercise before the test. The test will be conducted on a treadmill. A comfortable running speed acceptable to the participant will be set. The treadmill's incline will be increased by 10% every two minutes until the individual reaches their physical limit and can no longer continue. During this test, a respiratory mask and gas analyzer will be used to measure the concentration of oxygen (O2) and carbon dioxide (CO2) in the breath to calculate VO2max.
* Sample collection: Serum(vein blood extraction from the wrist or elbow by a nurse with a nursing qualification), feces, and urine
* Behaviour monitor: physical activity and food intake.

  * Physical activity：Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day with less than 12 hours of wear. For a valid measure the goal is to get 2 weekday and 2 weekend days.
  * Food intake：Photographic and food weighing methods to record food intake for two random days before intervention.

Exercise intervention:

* Exercise period: 12 weeks
* Exercise frequency: 5 times a week
* Exercise modality: Under the supervision of the researcher, participants will run on a treadmill
* Exercise intensity: 60% of VO2max (running speed and treadmill incline determined based on VO2max)
* Exercise energy expenditure: 150Kcal (Weeks 1-4, gradually increase to 150Kcal in the first two weeks), 250Kcal (Weeks 5-8), 350Kcal (Weeks 9-12), increasing monthly.
* Weight monitoring: Record participants' body weight changes during exercise without informing participants of the changes.
* Heart rate monitoring: Participants need to wear a 24-hour heart rate recorder every months during exercise intervention to monitor heart rate changes.
* VO2max testing: Due to physiological and psychological adaptability,exercise will increase VO2max. To ensure consistent exercise intensity and energy expenditure, VO2max testing will be conducted every four weeks to adjust the speed and duration of exercise for the following each four weeks.
* Blood sample collection: Fasting blood will be collected every four weeks.

Immediately measurement after 12 weeks'exercise intervention (same as pre-exercise intervention baseline measurement):

* Anthropometric measurements: body weight, height, and body composition.
* Metabolic measurements: blood pressure, glucose, heart rate, energy expenditure, and cardiovascular function.
* Sample collection: Serum, feces, and urine.
* Behaviour monitor: physical activity and food intake.

Follow-up measurement 8 weeks post-completion of the exercise intervention (same as pre-exercise intervention baseline measurement):

* Anthropometric measurements: body weight, height, and body composition
* Metabolic measurements: blood pressure, glucose, heart rate, energy expenditure, and cardiovascular function
* Sample collection: Serum, feces, and urine
* Behaviour monitor: physical activity and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals
* BMI ≥ 18.5 kg/m2

Exclusion Criteria:

* Individuals who have undergone major surgery in the past 6 months (excluding tooth extraction);
* Individuals on long-term medication;
* Individuals with metabolic and cardiovascular diseases such as diabetes, hypoglycemia, and hypertension;
* Individuals with exercise-related injuries, including joint diseases and fractures;
* Individuals diagnosed with infectious diseases such as HIV, tuberculosis, malaria, etc.;
* Individuals with mental and neurological disorders including anorexia nervosa;
* Individuals who have attempted weight loss or gain through various methods in the past three months;
* Individuals in preconception, pregnancy, and lactation periods;
* Individuals with autism and those with metal implants in their bodies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in TEE. | Three times, it takes 14 days for each time: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  The change in TEE will be evaluated using the DLW method before and after exercise intervention.
Change in TEF and REE. | Three times, it takes 1 days for each time: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  The change in BEE and TEF will be measured through indirect calorimetry in a respiratory chamber.
Change in exercise energy expenditure. | Three times, it takes 14 days for each time: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  The change in exercise energy expenditure will be assessed using indirect calorimetry with a respiratory hood system (COSMED).
Change in food intake. | Three times, food intake assessment takes 2 days: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  Food intake will be assessed using a 2-day food record complemented by photographing and weighing the food before and after consumption.
Change in physical activity. | Three times, it takes takes 14 days: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  The physical activity levels of the participants will be monitored through the use of a GT3X accelerometer.

SECONDARY OUTCOMES:
Change in fasting glucose and postprandial glucose. | Three times, 7 days per each time: before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  The continuous glucose monitoring system (Medtronic) will record the glucose concentration in mmol/L for 7 days.
Change in circulating hormones and metabolites. | 8 times, 1 minutes for each collection, 7 days for analysis. Every months (week0, 4, 8,12, and 30), and after exercise energy expenditure test(week 0,12, and 20))
  During the experiment, the nurse will collect the fasting blood sample in each month throughout exercise intervention, right after the first and last exercise session, and the 8 weeks upon completion of exercise intervention. Metabolomics will analyze the impact of an exercise intervention on metabolites.
Change in intestinal microbiota. | Three times, it takes 5 minutes for collection, 7 days for analysis. before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  Feces will be collected for gut microbiome analysis of intestinal microbiota.
Change in fat mass. | Three times, it takes 10 minutes, before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Change in fat free mass. | Three times, it takes 2 minutes for each time, before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, MC-980).
Change in bone mass. | Three times, it takes 7 minutes for each time, before exercise intervention (week 0), immediately after exercise intervention (week 12), and 8 weeks post-completion of exercise intervention (week 20).
  Bone mass will be measured by DXA( Horizon Wi, HOLOGIC)

OTHER OUTCOMES:
Change in metabolic energy expenditure before and after an intense exercise session. | 1 day, before and after the first intense exercise session
  Participants will enter the chamber at night to equilibrate the chamber air and become familiar with the setup. The initial light exposure day in the respiratory chamber, labeled as day 0, will not involve any exercise. The subsequent 24 hours will mark the beginning of the exercise intervention, designated as day 1. The alterations of BEE and TEF will be assessed using indirect calorimetry within the respiratory chamber between day 0 and day 1.
Change in metabolic energy expenditure upon completion of exercise intervention. | 1 day, before and after the last exercise session
  Participants will enter the chamber at the second last exercise intervention night to equilibrate the chamber air and become familiar with the setup. The initial light exposure day in the respiratory chamber, labeled as day 84, will be the last day of exercise intervention. The subsequent 24 hours will mark the first day of the completion of exercise intervention, designated as day 85. The alterations of BEE and TEF will be assessed using indirect calorimetry within the respiratory chamber between day 84 and day 85.

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences, Shenzhen, Guangdong, China

REFERENCES:
- [Result] Pontzer H, Durazo-Arvizu R, Dugas LR, Plange-Rhule J, Bovet P, Forrester TE, Lambert EV, Cooper RS, Schoeller DA, Luke A. Constrained Total Energy Expenditure and Metabolic Adaptation to Physical Activity in Adult Humans. Curr Biol. 2016 Feb 8;26(3):410-7. doi: 10.1016/j.cub.2015.12.046. Epub 2016 Jan 28. PMID 26832439
- [Result] Careau V, Halsey LG, Pontzer H, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Das SK, Cooper R, Dugas LR, Eaton SD, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reilly JJ, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Luke AH, Rood J, Sagayama H, Schoeller DA, Wong WW, Yamada Y, Speakman JR; IAEA DLW database group. Energy compensation and adiposity in humans. Curr Biol. 2021 Oct 25;31(20):4659-4666.e2. doi: 10.1016/j.cub.2021.08.016. Epub 2021 Aug 27. PMID 34453886
- [Result] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- See also: Constrained Total Energy Expenditure and Metabolic Adaptation to Physical Activity in Adult Humans — https://pubmed.ncbi.nlm.nih.gov/26832439/
- See also: Energy compensation and adiposity in humans — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8551017/
- See also: A standard calculation methodology for human doubly labeled water studies — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7897799/